CLINICAL TRIAL: NCT03831685
Title: Contribution of Pre-hospital Blood Lactate Level for Pre-hospital Orientation of Septic Shock
Brief Title: Blood Lactate Level for Pre-hospital Orientation of Septic Shock
Acronym: LAPHSUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: Fire Brigade Of Paris Emergency Medicine Dept (Other); University Hospital, Grenoble (Other); University Hospital, Toulouse (Other); University Hospital Center of Martinique (Other)
Responsible Party: Principal Investigator, Romain Jouffroy, PI, Hôpital Necker-Enfants Malades
Other Study IDs: LAPHSUS study
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Sepsis; Lactate Blood Increase
Keywords: sepsis; lactate; prehospital; prediction; mortality
MeSH Terms: conditions — Sepsis; Hyperlactatemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample — Patients meeting the inclusion criteria and none of the non-inclusion criteria will benefit from 2 venous blood samples in order to precise the initial blood lactate level, e.g. at the first medical contact, and the final blood lactate level, e.g. at the hospital admission.

SUMMARY:
In the pre-hospital setting, the severity assessment of septic shock is essential to decide the optimal initial in-hospital level of care. As clinical signs can be faulted, there is a need for an additional element in order to enhance the severity assessment and to decide in-hospital admission in the intensive care unit (ICU) or in the emergency department (ED). Point of care medical device yielding blood lactate levels since the pre-hospital setting may give an easy and valuable element for the severity assessment and the decision-making.

The aim of this study is to provide clinical evidence that the pre-hospital blood lactate level predicts the 30-day mortality of patients with septic shock.

DETAILED DESCRIPTION:
This trial is a prospective, observational, non-randomized controlled study. A total of 1000 patients requiring mobile intensive care unit intervention for a septic shock in the pre-hospital setting will be included. Pre-hospital blood lactate levels will not be taken into account to decide patients treatments and/or ED or ICU admission. In the pre-hospital setting, each patient will benefit from 2 measurements of blood lactate level: initial measurement at the first contact, and final measurement at the hospital admission with a specific point of care medical device.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years either sex
* Severe sepsis according to the French anesthesiology and intensive care society (SFAR) and intensive care society (SRLF) conference 2005 defined by the existence of an infectious disease and at least one the following:

  * Low blood pressure prior to volume expansion
  * Glasgow coma scale < 13
  * Skin mottling score > 2
* Septic shock according to the French anesthesiology and intensive care society (SFAR) and intensive care society (SRLF) conference 2005 definition

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Serious comorbid conditions with a not to be reanimated status known since pre-hospital setting
* Patients with guardianship or curator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock in the pre-hospital setting requiring mobile intensive care unit intervention
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Mortality after inclusion | 30 days
  mortality rate

SECONDARY OUTCOMES:
Intensive Care Unit length of stay | 90 days
  Duration of ICU length of stay
Hospital length of stay | 90 days
  Duration of Hospital length of stay
Mechanical ventilatory support | 30 days
  Duration of mechanical ventilation
Hemodynamic support | 30 days
  Duration of catecholamines' infusion
Duration of hemodiaflitration | 30 days
  Duration of extra renal support

CONTACTS AND LOCATIONS:
Overall Officials: Romain Jouffroy, MD, Principal Investigator — APHP - Necker enfants malades Hospital - SAMU Anesthesiology and intensive care unit
Locations (1):
- APHP Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marecaux G, Pinsky MR, Dupont E, Kahn RJ, Vincent JL. Blood lactate levels are better prognostic indicators than TNF and IL-6 levels in patients with septic shock. Intensive Care Med. 1996 May;22(5):404-8. doi: 10.1007/BF01712155. PMID 8796390
- [Background] Bakker J, Coffernils M, Leon M, Gris P, Vincent JL. Blood lactate levels are superior to oxygen-derived variables in predicting outcome in human septic shock. Chest. 1991 Apr;99(4):956-62. doi: 10.1378/chest.99.4.956. PMID 2009802
- [Background] Cicarelli DD, Vieira JE, Bensenor FE. [Lactate as a predictor of mortality and multiple organ failure in patients with the systemic inflammatory response syndrome.]. Rev Bras Anestesiol. 2007 Dec;57(6):630-8. doi: 10.1590/s0034-70942007000600005. Portuguese. PMID 19462139
- [Background] Gaieski DF, Goyal M. Serum lactate as a predictor of mortality in emergency department patients with infection: does the lactate level tell the whole story? Ann Emerg Med. 2005 Dec;46(6):561-2; author reply 562. doi: 10.1016/j.annemergmed.2005.07.021. No abstract available. PMID 16308078
- [Background] Mikkelsen ME, Miltiades AN, Gaieski DF, Goyal M, Fuchs BD, Shah CV, Bellamy SL, Christie JD. Serum lactate is associated with mortality in severe sepsis independent of organ failure and shock. Crit Care Med. 2009 May;37(5):1670-7. doi: 10.1097/CCM.0b013e31819fcf68. PMID 19325467
- [Background] Shapiro NI, Howell MD, Talmor D, Nathanson LA, Lisbon A, Wolfe RE, Weiss JW. Serum lactate as a predictor of mortality in emergency department patients with infection. Ann Emerg Med. 2005 May;45(5):524-8. doi: 10.1016/j.annemergmed.2004.12.006. PMID 15855951
- [Background] Arnold RC, Shapiro NI, Jones AE, Schorr C, Pope J, Casner E, Parrillo JE, Dellinger RP, Trzeciak S; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Multicenter study of early lactate clearance as a determinant of survival in patients with presumed sepsis. Shock. 2009 Jul;32(1):35-9. doi: 10.1097/shk.0b013e3181971d47. PMID 19533847